CLINICAL TRIAL: NCT06689943
Title: Pain After Strabismus Surgery: Post-Operative Outcomes Using Courses of Acetaminophen in Children
Brief Title: Pain After Strabismus Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Hawke H. Yoon, Attending Ophthalmologist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-7067
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Strabismus
Keywords: pain; strabismus surgery
MeSH Terms: conditions — Strabismus; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tylenol as needed (Active Comparator): Tylenol prescribed to be taken as needed for pain management for 48 hours after surgery
  Interventions: Drug: Tylenol
- Tylenol every 6hrs (Experimental): Tylenol prescribed to be taken very 6 hours for pain management for 48 hours after surgery
  Interventions: Drug: Tylenol

INTERVENTIONS:
Drug: Tylenol — Tylenol for children
  Other Names: acetaminophen

SUMMARY:
At Ann & Robert H. Lurie Children's Hospital of Chicago (Lurie Children's), the current practice is to prescribe children with oral Tylenol as needed every 4-6 hours post strabismus surgery. Prescribing Tylenol "as needed" leaves more room for error for parents to be under-dosing their children, which can lead to avoidable pain. This study aims to figure out if children ages 4-12 years old will feel significantly less pain and discomfort when given regimented Tylenol every 6 hours for 48 hours after strabismus surgery (eye muscle surgery) compared to controls whose parents are instructed to give Tylenol every 4-6 hours as needed for 48 hours after surgery. To date, there have been no studies comparing patient outcomes between those taking Tylenol regimen and those receiving Tylenol as needed after pediatric surgery.

DETAILED DESCRIPTION:
Main hypothesis:

Children ages 4-12 years will feel significantly less pain and discomfort when given regimented Tylenol every 6 hours for 48 hours after strabismus surgery (surgery to correct misaligned eyes) compared to controls whose parents are instructed to give Tylenol every 4-6 hours as needed for 48 hours after surgery.

Primary Objective At Lurie Children's, the current standard practice is for patients to be prescribed oral acetaminophen as needed every 4-6 hours after strabismus surgery. However, making the acetaminophen "as needed" leaves room for error for parents to be underdosing their children and, thus, leads to increased pain felt by these pediatric patients. To date, there have been no studies comparing patient satisfaction outcomes between a group taking a course of scheduled acetaminophen every 6 hours and to a group instructed to take as needed. The investigators plan to study the differences between these two groups by using the Parent's Post-operative Pain Measure (PPPM) questionnaire to survey parents and the Faces Pain Scale-Revised to survey children at their post-operative appointment.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4-12 years old
* Children receiving single muscle, bilateral horizontal strabismus surgery (that is, children who are having only one horizontal eye muscle in each eye operated on) at Lurie Children's hospital in Chicago, IL
* ASA classification 1 or 2. Note: ASA is a physical status classification system (scale of 1-6) created by the American Society of Anesthesiologists to describe patients prior to surgery. ASA 1 or 2 means the patient is either healthy or has mild systemic disease prior to surgery.

Exclusion Criteria:

* ASA classification 3 or higher (patient has severe systemic disease or worse)
* Contraindication to toradol (anesthesia)
* Contraindication to acetaminophen
* Previous strabismus surgery

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent reported Pain score using the Parent's Post-operative Pain Measure | From enrollment to 1 day after surgery
  Pain score reported by parent validated questionnaire- Scale from 0 to 29, 0 is no pain and 29 is the worst pain.
Child reported pain score using the Faces Pain Scale- Revised | 2-4 days after surgery
  Child reported pain using Faces Pain Scale revised questionnaire. Scale from 0 to 5; 0 is no pain and 5 is the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walther-Larsen S, Aagaard GB, Friis SM, Petersen T, Moller-Sonnergaard J, Romsing J. Structured intervention for management of pain following day surgery in children. Paediatr Anaesth. 2016 Feb;26(2):151-7. doi: 10.1111/pan.12811. Epub 2015 Nov 12. PMID 26559643
- [Background] Vons KM, Bijker JB, Verwijs EW, Majoor MH, de Graaff JC. Postoperative pain during the first week after adenoidectomy and guillotine adenotonsillectomy in children. Paediatr Anaesth. 2014 May;24(5):476-82. doi: 10.1111/pan.12383. Epub 2014 Mar 20. PMID 24646093
- [Background] Ghai B, Makkar JK, Wig J. Postoperative pain assessment in preverbal children and children with cognitive impairment. Paediatr Anaesth. 2008 Jun;18(6):462-77. doi: 10.1111/j.1460-9592.2008.02433.x. Epub 2008 Mar 18. PMID 18363630
- [Background] de Azevedo CB, Carenzi LR, de Queiroz DL, Anselmo-Lima WT, Valera FC, Tamashiro E. Clinical utility of PPPM and FPS-R to quantify post-tonsillectomy pain in children. Int J Pediatr Otorhinolaryngol. 2014 Feb;78(2):296-9. doi: 10.1016/j.ijporl.2013.11.027. Epub 2013 Dec 1. PMID 24370467
- [Background] Chambers CT, Reid GJ, McGrath PJ, Finley GA. Development and preliminary validation of a postoperative pain measure for parents. Pain. 1996 Dec;68(2-3):307-13. doi: 10.1016/s0304-3959(96)03209-5. PMID 9121819
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704